CLINICAL TRIAL: NCT06787508
Title: Exploration of Repeated High-frequency Transcranial Magnetic Stimulation for the Treatment of Acute Phase Aphasia in Post-stroke Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Fei Xiao, professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-335-01
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Aphasia; Control Patients
Keywords: Post stroke aphasia; TMS
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Adopting double-blind method: 1) Patients do not know which group they are assigned to; 2) Physicians who group patients do not perform scale scoring and are only responsible for analyzing data before and after treatment; 3) Other neurologists who do not know the specific grouping will perform scale scoring and TMS treatment on patients before and after treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Targeting the left M1 area, continuous high-frequency stimulation was performed at a frequency of 10Hz with 80-100% TEP for 5 minutes each time, twice a day for a total of 5 days
  Interventions: Device: TMS
- Control group (Sham Comparator): Consistent with the experimental group protocol, the magnetic stimulation probe is a false stimulation probe, which only produces sound but does not actually produce stimulation
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Continuous high-frequency transcranial magnetic stimulation therapy Targeting the left M1 area, continuous high-frequency stimulation was performed at a frequency of 10Hz with 80-100% TEP for 5 minutes each time, twice a day for a total of 5 days
  Arms: Test group
Device: TMS — Consistent with the experimental group protocol, the magnetic stimulation probe is a false stimulation probe that only produces sound but does not actually produce stimulation
  Arms: Control group

SUMMARY:
Stroke is currently an important cause of death and disability among adults worldwide, with acute ischemic stroke being the most common type of stroke, accounting for 69.6% -72.8% of new strokes in China. The time division of the acute phase generally refers to the onset time within 1-2 weeks. About 21-38% of stroke patients have post-stroke aphasia. Post stroke aphasia is usually an acquired language disorder caused by damage to the language functional areas of the dominant hemisphere, characterized by varying degrees of impairment in some or all language functions, including speaking, listening and understanding, paraphrasing, naming, reading, and calligraphy abilities. Rehabilitation treatment for cerebral infarction should be done early rather than late. Based on this, this study aims to explore transcranial magnetic stimulation therapy for post-stroke aphasia patients in the acute phase. By regulating the balance of cortical excitability on both sides of the healthy and affected areas, early speech function rehabilitation can be achieved, which is necessary for improving the quality of life of post-stroke aphasia patients

DETAILED DESCRIPTION:
Post stroke aphasia (PSA) is an acquired communication disorder caused by brain injury, characterized by various functional impairments such as self speech, repetition, naming, auditory comprehension, reading, and writing. PSA is one of the serious sequelae of stroke, which seriously affects the quality of life of patients. Early intervention in speech therapy can to some extent restore patients' functional communication abilities. Transcranial magnetic stimulation (TMS) is currently the most widely used non-invasive therapy. TMS can generate a magnetic field through the principle of magnetoelectric conversion, which can penetrate the skull and generate a super threshold current, allowing neurons in the target brain area to discharge. High frequency rTMS (generally frequency>5HZ) is usually applied to the affected side, aiming to improve aphasia symptoms by directly promoting the excitability of the affected cortex.

The rehabilitation treatment for PSA patients often stabilizes within a few months after stroke, and early intervention may maximize potential benefits. At present, research on high-frequency rTMS is mostly limited to the subacute or chronic phase. Therefore, this study aims to explore a safe and effective TMS treatment method during the acute phase.

ELIGIBILITY:
Inclusion Criteria:1) Age ≥ 18 years old 2) Head MR confirms new onset of cerebral infarction, and aphasia symptoms are caused by cerebral infarction 3) Patient's hospitalization history is within 7 days 4) Can cooperate to complete all required inspection items and scales 5) Sign informed consent form 6) Right handed -

Exclusion Criteria:1)Patients with aphasia caused by non cerebral infarction,2) Non acute phase cerebral infarction patients with a course of more than 7 days 3) Severe neurological disorders other than stroke, such as epilepsy and hemorrhagic stroke, are combined 4) Patients with poor general condition and unable to complete relevant examinations and scale scores, such as patients with malignant arrhythmia, tumor, severe infection, malignant hypertension, diabetes hyperosmolar coma, etc 5) Previous or current comorbidities of severe mental illnesses, such as depression, schizophrenia, etc 6) Patients who have previously or currently taken sedatives or large amounts of sleep aids 7) Contraindications for combined transcranial magnetic stimulation: presence of metal or other implants (such as pacemakers) in the body 8) Pregnancy and lactation period

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
BDAE Scale Score | From before treatment to 1 month after treatment, a total of 3 time points
  Collect the scores of the experimental group/control group on the Aphasia Scale before and after treatment, calculate the difference in scores for each patient and the average value of each component. Assuming that the average difference between groups is greater than 20%, it is considered that there is a significant difference

SECONDARY OUTCOMES:
Electrophysiological measurement | From before treatment to 1 month after treatment, a total of 3 time points
  By collecting EEG/TMS data from patients, evaluate their electrophysiological characteristics and related changes at three time points from before treatment to one month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xiao, Professor, Study Director — First Affiliated Hospital of Chongqing Medical University; Jing Luo, associate professor, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Municipality Directly Under the Central Government, China

IPD SHARING:
Plan to Share IPD: Yes
With the consent of both researchers and participants, the original data can be obtained by contacting with the corresponding member.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2024.12~2025.06
Access Criteria: After obtaining informed consent from the patients and ensuring compliance with ethical principles, this study uses Case Report Forms (CRF) and questionnaires to collect subject information. The CRFs and questionnaires are stored in both paper and electronic databases. Data collection occurs after obtaining patients' informed consent at the time of their participation in the study assessment. Two members of the research team independently enter CRF data into the electronic database, and any discrepancies are reconciled before making changes to the entry. Original paper and electronic data are registered and stored in our department's clinical trial archive cabinet.